CLINICAL TRIAL: NCT03808740
Title: Orthostatic Intolerance After Bariatric Surgery
Acronym: RYGB
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to COVID-19 pandemic, recruitment was stopped. All the weight loss surgeries were stopped.. Weight Loss clinic (VWL) was closed for IN person visits. We could not recruit any participant for Non surgical weight loss category.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, MD, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 180499
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-06

CONDITIONS: Orthostatic Intolerance
MeSH Terms: conditions — Orthostatic Intolerance | interventions — Atomoxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Roux-en-Y gastric bypass (RYGB)/Atomoxetine (Experimental): Participants with standard of care RYGB will receive atomoxetine, 0.5 mg/kg/day for 3 days
  Interventions: Drug: Atomoxetine
- Vertical sleeve gastrectomy (VSG) /Atomoxetine (Experimental): Participants with standard of care VSG will receive atomoxetine 0.5 mg/kg/day for 3 days
  Interventions: Drug: Atomoxetine
- Roux-en-Y gastric bypass (RYGB)/Placebo (Placebo Comparator): Participants with standard of care RYGB will receive placebo 0.5 mg/kg/day for 3 days
  Interventions: Drug: Placebo
- Vertical sleeve gastrectomy (VSG)/ Placebo (Placebo Comparator): Participants with standard of care VSG will receive placebo 0.5 mg/kg/day for 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — atomoxetine 0.5 mg/kg/day.
  Other Names: strattera
  Arms: Roux-en-Y gastric bypass (RYGB)/Atomoxetine; Vertical sleeve gastrectomy (VSG) /Atomoxetine
Drug: Placebo — sugar pill
  Other Names: sugar pill
  Arms: Roux-en-Y gastric bypass (RYGB)/Placebo; Vertical sleeve gastrectomy (VSG)/ Placebo

SUMMARY:
More than 78 million adults in the U.S. are obese. Bariatric surgery is the only modality that results in sustained weight loss along with reversal of diabetes mellitus, and a decrease in cardiovascular events. Obesity is associated with increased sympathetic nervous system (SNS) activity that contributes to blood pressure regulation; sympathetic vasoconstrictor activity is maximally activated upon standing and is fundamental for the maintenance of orthostatic tolerance. After bariatric surgery, there is a significant and sustained reduction in SNS activity at three and six months after the procedure, which is related to weight loss. Recently, multiple retrospective studies have reported an orthostatic intolerance (OI) syndrome after bariatric surgery characterized by chronic pre-syncopal symptoms, syncope and orthostatic hypotension. In the Vanderbilt University Medical Center bariatric surgical center, 741 post-bariatric surgery patients reported OI symptoms, 98 (13.2%) of these patients, progressed to chronic OI and in17 cases, the OI was so disabling that patients initiated treatment with pressor agents. More than 50% of OI cases in the cohort developed the condition during a weight-stable period. Hence, investigators propose the novel hypothesis that after bariatric surgery, the persistent reduction in SNS activity contributes to impaired orthostatic tolerance, which is independent of weight loss.

DETAILED DESCRIPTION:
Considering that SNS vasoconstrictor activity depends on synaptic norepinephrine concentrations, investigators propose a proof-of-concept study to test the hypothesis that the norepinephrine transporter (NET) inhibitor, atomoxetine, which increases synaptic norepinephrine concentrations, will improve post-bariatric OI. Understanding the changes in SNS activity and its contribution to orthostatic tolerance after bariatric surgery is of utmost importance to unravel the mechanisms of a novel and unrecognized syndrome, post-bariatric OI. In 2014, nearly 200,000 individuals in the US underwent bariatric surgery, and the number of bariatric surgery procedures is expected to increase by 22% each year. It is projected, therefore, an increase in the incidence of post-bariatric OI.

Participants with Roux-en-Y gastric bypass (RYGB) and Vertical sleeve gastrectomy (VSG) will be studied.

OI is a chronic and disabling condition; treatment is challenging because current therapies have debatable efficacy.

The proposed application will not only provide central knowledge on the pathophysiology of this new syndrome but also will fill an unmet therapeutic need by repurposing NET inhibitors for the treatment of OI.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects that will undergo bariatric surgery or medical weight loss.
* Age 18-60 years
* BMI >35 kg/m2
* Weight < 400 lbs

Exclusion Criteria:

* Diabetes type 1
* Use of an alpha blockers, clonidine, beta-blockers.
* Pregnancy or breast-feeding. Women of childbearing potential will be required to have undergone tubal ligation or to be using an oral contraceptive or barrier methods of birth control.
* The use of any strong CYP2D6 inhibitor (e.g., fluoxetine, paroxetine, quinidine, tipranavir).
* Use of selective NET inhibitors.
* Use of monoamine oxidase inhibitors.
* Cardiovascular disease such as myocardial infarction within six months prior to the study, presence of angina pectoris, significant arrhythmia, congestive heart failure (left ventricular hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
* History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack
* Hematocrit < 34%
* Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
* Mental conditions rendering a subject unable to understand the nature, scope and possible consequences of the study
* Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, unlikelihood of completing the study, and investigator discretion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya Shiabao, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Cyndya Shibao, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 morbid obese patients, scheduled for bariatric surgery, were enrolled in this study.
  10 patients completed all 4 visits, which include a pre-surgical visit, a visit after 10% weight loss, and a visit after 3-months post-surgery. The demographic characteristics of these patients are shown in the table below.
  We could not enroll any patients, in Medical Weight loss category
Groups:
- Baseline (Pre-surgery, RYGB/VSG): Participants underwent Bariatic surgery Roux-en-Y gastric bypass (RYGB) / Vertical sleeve gastrectomy (VSG) for weight loss .
- Baseline Pre-hypocaloric Diet (Medical Weight Loss): Participants who underwent standard medical weight loss from the Vanderbilt Center for Weight Loss (VWL)
Period: Overall Study
Arm/Group | Baseline (Pre-surgery, RYGB/VSG) | Baseline Pre-hypocaloric Diet (Medical Weight Loss)
Started | 10 | 0
Completed | 10 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to COVID-19 pandemic, recruitment was stopped, all the weight loss surgeries and non-essential procedures, were stopped. Due to high COVID -19 prevalence the Vanderbilt Weight Loss clinic (VWL) was closed for IN person visits. We could not recruit any participant for Non surgical weight loss category.
Groups:
- Baseline Characteristics Before Participants Underwent Bariatric Surgery for Weight Loss: Participants underwent Bariatic surgery Roux-en-Y gastric bypass (RYGB) / Vertical sleeve gastrectomy (VSG) for weight loss .
- Baseline of Participants Before They Underwent Non Surgical (Medical) Weight Loss Program: Participants who underwent standard medical weight loss from the Vanderbilt Center for Weight Loss (VWL)
- Total: Total of all reporting groups
Arm/Group | Baseline Characteristics Before Participants Underwent Bariatric Surgery for Weight Loss | Baseline of Participants Before They Underwent Non Surgical (Medical) Weight Loss Program | Total
Number analyzed (Participants) | 10 | 0 | 10
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 42 (9.3) |  | 42 (9.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 9 | 0 | 9
  Gender: Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 166 (8.6) |  | 166 (8.6)
Fat Mass [Mean (Standard Deviation); unit: Kg] | 73 (12.18) |  | 73 (12.18)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m2] | 51 (8.27) |  | 51 (8.27)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm of Hg] | 128 (3.69) |  | 128 (3.69)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm of Hg] | 85 (4.69) |  | 85 (4.69)
Heart rate [Mean (Standard Deviation); unit: beats per minute] | 93 (7.93) |  | 93 (7.93)
Bariatric surgery type [Count of Participants; unit: Participants]
  Roux-en-Y Gastric By-Pass procedures | 7 |  | 7
  Vertical Sleeve Gastric By-Pass | 3 |  | 3
Total Blood Volume [Mean (Standard Deviation); unit: Litres] | 316.1 (6) |  | 316.1 (6)
Red Blood Cell volume [Mean (Standard Deviation); unit: ml] | 1973 (136.5) |  | 1973 (136.5)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Measurements During Orthostatic Challenge With a Head up Tilt (HUT at 60 Degrees) Before and After Bariatric Surgery: at 2 Timepoints: After 10% Weight Loss and After 3 Months
Description: To assess the hemodynamic (Blood Pressure) changes during an orthostatic challenge with a head up tilt (HUT at 60 degrees) before and after bariatric surgery, at two time-points: after 10% weight loss (10% WL) and after 3 months, in morbidly obese patients.
  Our primary endpoint (orthostatic tolerance, OT) is defined as the time between the start of the 60 degree HUT until pre-syncope Orthostatic hemodynamics were analyzed as the area under the curve (AUC) after baseline-correction during HUT.
Time Frame: 0- 3 months
Population: Orthostatic hemodynamics (SBP, DBP, HR) were analyzed as the area under the curve (AUC) after baseline-correction during HUT
Measure: Mean (Standard Deviation); unit: mmHg*hr
Groups:
- Pre- Bariatric Participants: Parameters taken before the subject underwent any of the Bariatric surgery Roux-en-Y gastric bypass (RYGB) / Vertical sleeve gastrectomy (VSG) were analysed for Orthostatic tolerance. .
- Participants After 10% of Weight Loss: Participants who underwent Bariatic surgery Roux-en-Y gastric bypass (RYGB) / Vertical sleeve gastrectomy (VSG) were analyzed for Orthostatic tolerance after 10% of weight loss in morbidly obese patients
- Participants After 3 Months of the Surgery: Participants who underwent Bariatic surgery Roux-en-Y gastric bypass (RYGB) / Vertical sleeve gastrectomy (VSG) were analyzed for Orthostatic tolerance after 3 months in morbidly obese patients
Arm/Group | Pre- Bariatric Participants | Participants After 10% of Weight Loss | Participants After 3 Months of the Surgery
Number analyzed (Participants) | 10 | 10 | 10
mmHg*hr
  Systolic Blood pressure: analyze as Area under the curve (AUC) after baseline-correction during HUT. | 113 (72.41) | 56.02 (30.68) | 39.4 (28.53)
  Diastolic Blood pressure:analyze as Area under the curve (AUC) after baseline-correction during HUT | 303.7 (93.74) | 60.98 (29.54) | 39.44 (28.53)

2. Primary Outcome: Cardiac Output During Orthostatic Challenge With a Head up Tilt (HUT at 60 Degrees) Before and After Bariatric Surgery: at 2 Timepoints: After 10% Weight Loss and After 3 Months
Description: To assess the hemodynamic (cardiac output [CO]) and cardiovascular autonomic changes during an orthostatic challenge with a head up tilt (HUT at 60 degrees) before and after bariatric surgery, at two time-points: after 10% weight loss (10% WL) and after 3 months, in morbidly obese patients.
  Our primary endpoint (orthostatic tolerance, OT) is defined as the time between the start of the 60 degree HUT until pre-syncope Orthostatic hemodynamics were analyzed as the area under the curve (AUC) after baseline-correction during HUT.
Time Frame: 0- 3 months
Population: Orthostatic hemodynamics (Cardiac Output ) were analyzed as the area under the curve (AUC) after baseline-correction during HUT
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Pre- Bariatric Participants | Participants After 10% of Weight Loss | Participants After 3 Months of the Surgery
Number analyzed (Participants) | 10 | 10 | 10
L/min | 9.124 (8.066) | 3.562 (2.522) | 4.916 (3.652)

3. Primary Outcome: Stroke Volume Measurements During Orthostatic Challenge With a Head up Tilt (HUT at 60 Degrees) Before and After Bariatric Surgery: at 2 Timepoints: After 10% Weight Loss and After 3 Months
Description: To assess the hemodynamic (stroke volume [SV]) and cardiovascular autonomic changes during an orthostatic challenge with a head up tilt (HUT at 60 degrees) before and after bariatric surgery, at two time-points: after 10% weight loss (10% WL) and after 3 months, in morbidly obese patients.
  Our primary endpoint (orthostatic tolerance, OT) is defined as the time between the start of the 60 degree HUT until pre-syncope Orthostatic hemodynamics were analyzed as the area under the curve (AUC) after baseline-correction during HUT.
Time Frame: 0- 3 months
Population: Orthostatic hemodynamics (Stroke volume) were analyzed as the area under the curve (AUC) after baseline-correction during HUT
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Pre- Bariatric Participants | Participants After 10% of Weight Loss | Participants After 3 Months of the Surgery
Number analyzed (Participants) | 10 | 10 | 10
mL | 116.2 (56.5) | 148 (78.61) | 105.6 (60.04)

4. Primary Outcome: Calculated Total Peripheral Resistance During Orthostatic Challenge With a Head up Tilt (HUT at 60 Degrees) Before and After Bariatric Surgery: at 2 Timepoints: After 10% Weight Loss and After 3 Months
Description: To assess the hemodynamic ( total peripheral resistance [TPR]) and cardiovascular autonomic changes during an orthostatic challenge with a head up tilt (HUT at 60 degrees) before and after bariatric surgery, at two time-points: after 10% weight loss (10% WL) and after 3 months, in morbidly obese patients.
  Our primary endpoint (orthostatic tolerance, OT) is defined as the time between the start of the 60 degree HUT until pre-syncope
Time Frame: 0- 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg*L/min
Arm/Group | Pre- Bariatric Participants | Participants After 10% of Weight Loss | Participants After 3 Months of the Surgery
Number analyzed (Participants) | 10 | 10 | 10
mmHg*L/min | 9.162 (5.995) | 7.239 (6.245) | 9.167 (4.458)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Due to high COVID -19 prevalence the Vanderbilt Weight Loss clinic (VWL) was closed for IN person visits. We could not recruit any participant for Non surgical -Medical weight loss category.
Groups:
- Baseline (Pre-surgery, RYGB/VSG): Participants underwent Bariatic surgery Roux-en-Y gastric bypass (RYGB) / Vertical sleeve gastrectomy (VSG) for weight loss .
  Participants in this group were randomized in 1:1 ratio with Atomoxetine 0.5mg/kg/day for 3 days OR Placebo
Arm/Group | Baseline (Pre-surgery, RYGB/VSG) | Baseline Pre-hypocaloric Diet (Medical Weight Loss)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT03808740/Prot_SAP_000.pdf